CLINICAL TRIAL: NCT00253201
Title: Efficacy, Tolerability and Safety of Galantamine in the Treatment of Alzheimer's Disease
Brief Title: A Study of the Safety and Effectiveness of Two Doses of Galantamine Versus Placebo in the Treatment of Patients With Alzheimer's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR006025
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2010-11

CONDITIONS: Alzheimer Disease; Dementia
Keywords: Alzheimer's disease; dementia; brain disease; memory loss; galantamine; placebo; caregiver; quality of life; resource utilization
MeSH Terms: conditions — Alzheimer Disease; Dementia; Brain Diseases; Memory Disorders | interventions — Galantamine

INTERVENTIONS:
Drug: galantamine hydrobromide

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of two doses of galantamine (a drug for treating dementia) versus placebo in the treatment of patients with Alzheimer's disease.

DETAILED DESCRIPTION:
Dementia is a chronic, progressive brain disease that may involve a number of symptoms, including memory loss and changes in personality, behavior, judgment, attention span, language and thought. The most common type of dementia is Alzheimer's disease. Over time, patients with Alzheimer's disease may lose ability to perform daily tasks related to personal care (for example, bathing, dressing, and eating) and may be unable to handle money or travel to familiar places. Several small clinical trials have shown galantamine to be safe and effective in treating the symptoms associated with Alzheimer's disease. Doses studied have ranged from 15 - 60 mg/day, with galantamine administered two or three times daily. Additional information is needed to determine the optimal dose regimen for galantamine in the treatment of Alzheimer's disease. This multicenter, double-blind, placebo-controlled study evaluates the safety and effectiveness of two doses of galantamine, each given twice daily, in the treatment of patients with Alzheimer's disease. All patients initially receive placebo for a 1-month period and then receive one of two doses of galantamine (beginning with 4 mg twice daily and gradually increasing to 12 or 16 mg twice daily) or placebo for 6 months. The primary measures of effectiveness include the change from baseline to the end of treatment in the ADAS-cog/11 score (Alzheimer's Disease Assessment Scale: sum of 11 cognitive items) and the CIBIC-plus (Clinician's Interview Based Impression of Change - Plus Caregiver Input) score. Additional measures of effectiveness assessed at the end of the treatment include the ADAS-cog/13 score (Alzheimer's Disease Assessment Scale: sum of 13 cognitive items) and the Disability Assessment for Dementia (DAD) score. Safety evaluations (incidence of adverse events, electrocardiograms (ECGs), physical examinations, laboratory tests) are performed throughout the study. Caregiver quality of life (Psychological General Well Being Index, (PGWB)) and health/social care resource utilization (physician and other health care professional visits, use of social services, etc.) is also assessed throughout the study by questionnaires answered by the caregivers. Blood samples are taken throughout the study to determine the concentration of drug in the blood. Patients may participate in an optional portion of the study in which their genetic material is analyzed to see if contains something that would affect the way galantamine is used by their bodies. The study hypothesis is that galantamine administered in either dose is effective in the treatment of Alzheimer's disease as compared with placebo, and is well tolerated. This study will be conducted in the United States. A companion study of exact design will be conducted internationally. Galantamine, 12 or 16 mg tablets (or placebo), by mouth twice daily for 6 months, beginning with 4 mg twice daily and gradually increasing to 12 or 16 mg twice daily.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients with a diagnosis of Alzheimer's disease according to the National Institute of Neurological and Communicative Disorders and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria (including patients living independently in residential homes for the elderly or day patients)
* have mild to moderate dementia, as evidenced by a Mini-Mental Status Examination (MMSE) score of 11 - 24, and a score of at least 12 on the cognitive portion of the Alzheimer's Disease Assessment scale (ADAS-cog)
* history of at least a 6 months of gradual and progressive cognitive decline
* have a consistent informant to accompany the patient on scheduled visits

Exclusion Criteria:

* Neurogenerative disorders such as Parkinson's disease
* dementia caused by small strokes or cerebrovascular disease
* cognitive impairment resulting from acute cerebral trauma, cerebral damage due to a lack of oxygen, vitamin deficiency, infections such as meningitis or AIDS, significant endocrine or metabolic disease, mental retardation, or a brain tumor
* having epilepsy, significant psychiatric disease, active peptic ulcer, clinically significant liver, kidney or lung disorders, or heart disease
* females of child bearing potential without adequate contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 636 (Actual)
Dates: Study Completion 1997-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline to the end of treatment in ADAS-cog/11 (Alzheimer's Disease Assessment Scale: sum of 11 cognitive items) and CIBIC-plus (Clinician's Interview Based Impression of Change - Plus Caregiver Input) scores

SECONDARY OUTCOMES:
Change from baseline to the end of treatment in ADAS-cog/13 and DAD scores; Concentration of drug in blood; PGWB; Health/social care resource use; Incidence of adverse events; Changes in laboratory tests, ECGs and physical examinations

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- [Result] Raskind MA, Peskind ER, Wessel T, Yuan W. Galantamine in AD: A 6-month randomized, placebo-controlled trial with a 6-month extension. The Galantamine USA-1 Study Group. Neurology. 2000 Jun 27;54(12):2261-8. doi: 10.1212/wnl.54.12.2261. PMID 10881250
- [Result] Raskind MA, Peskind ER, Truyen L, Kershaw P, Damaraju CV. The cognitive benefits of galantamine are sustained for at least 36 months: a long-term extension trial. Arch Neurol. 2004 Feb;61(2):252-6. doi: 10.1001/archneur.61.2.252. PMID 14967774
- See also: A study of the safety and effectiveness of 2 doses of galantamine in patients with Alzheimer's disease — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=699&filename=CR006025_CSR.pdf